CLINICAL TRIAL: NCT02791607
Title: Technical Development of P16-INk4A-expressing Circulating Tumor Cells Detection Comparing With Human Papillomavirus Infection in Cancer Tissue in Patients With Head and Neck Cancer and Its Clinical Relevance.
Brief Title: The Clinical Relevance of P16 Expressing CTCs Detection Comparing With HPV Infection in Cancer Tissue in HNSCC Patients.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jason Chia-Hsun Hsieh, Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Other Study IDs: CTCHNSCC03; CMRPG3E1631-1633 (Other: Grantor or Funder CMRPG3E1631-1633)
Record Dates: First submitted 2016-06-01; First posted 2016-06-07 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Recurrence; Metastasis; Death
Keywords: Circulating tumor cells; Head and neck cancer; Survival Prognosis; P16Ink4A; HPV
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis; Death; Neoplastic Cells, Circulating; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: None Retained — Blood samples were drawn by standard procedure, stored in EDTA-coating tubes in 4 degree temperature, then sent for CTCs counting and analysis.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
HNSCC is the 4th highest incidence of cancer and 6th of cancer death of the males in Taiwan. Because the patients were mainly middle-aged male, the disease eventually resulted in a huge loss of labor force, productivity and a huge burden of family supports and medicinal costs. Currently, the primary treatments of HNSCC are mainly surgery, radiotherapy, chemotherapy or targeted therapy or concurrent chemoradiotherapy. Compared to oral cavity cancer, patients with pharyngeal cancer would possibly harbor HPV infections and have better treatment outcomes, prognosis and survival with clinically significance; however, the investigator's reports showed quite the opposite prognostic value in oral cavity cancer. The inconsistent data urges us to investigate further. Fortunately, in recent years, The investigator have developed a new method for isolation and detection of CTCs in HNSCC patients.The investigator's data found that high level of CTCs in patients with HNSCC and might be associated with disease prognosis, response to treatment and distant metastasis. This novel tool enhances the studies addressing on metastases or recurrence process in HNSCC patients. However, the investigator did not focus whether if the dynamic change of CTCs and specific surface markers on CTCs, such as P16+ CTCs are clinically meaningful.

Therefore, in the first year, the investigator will utilize the investigator's developing device and protocol to isolate high-purity CTCs to further identify P16+ on CTCs. In the following 2 years of the project, the investigator will enroll 150 freshly diagnosed patients with oral cavity, oropharyngeal, hypopharyngeal and laryngeal cancer at all stages (75 P16+ and 75 P16- patients) and 30 healthy donors for cell line tests, and then analyze CTCs, background white blood cells signals, and their initial biopsied tissue for P16 positivity test. Further statistical tests with clinical conditions (disease status, treatment effects, progression or distant metastasis and death) will be performed to elucidate their clinical significance.Hopefully, the investigator will clarify the clinical significance of circulating P16 expression status on CTCs by this study and provide a new biomarker for clinical cancer care.

DETAILED DESCRIPTION:
1. Establish a protocol and a practical platform to longitudinally isolate, enumerate CTCs in patients with HPV+-head and neck cancer during the treatment course.
2. Elucidate the clinical significance of P16 INK4A -expressing CTCs to cancer status and treatment response.
3. Verify that dynamically monitoring P16 status and changes during anti-cancer treatment is feasible and clinically meaningful to survival or treatment responses.
4. Analyze different habitual conditions, i.e. alcohol, cigarette and betel nut use to P16-expressing CTCs.
5. Establish a good model to follow-up a specific surface marker on CTCs, which could be possibly utilized in other cancers with their particular markers (i.e. CEA on gastric cancer, Her2 on breast cancer)

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytopathologically proven head and neck squamous cell carcinoma Age ≥ 20 years. Measurable or evaluable disease according to Response Evaluation Criteria In Solid Tumors(RECIST) criteria.

Ability to sign informed consent.

Exclusion Criteria:

* Prior cancers within 5 years, except for non-melanoma skin cancers, and in situ cervical cancers.

Inability to completely with study and/or follow-up procedures.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in three branch hospitals of Chang Gung Memorial Hospital, Taiwan including Keelung, Linkou, Taipei. Locally advanced or recurrent/metastatic head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | one year
  Measure response or progression events via all available imaging studies, including Chest-Xray, CT scans, or MRI, PET study. The relationship between CTCs number and time from CTCs checkpoint to disease progression will be analyzed.

SECONDARY OUTCOMES:
Overall survival | one year
  All causes of death would be documented and the relationship between CTCs number and time from CTCs checkpoint to death will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hsun Hsieh, M.D, M.S, Principal Investigator — Division of Hematology-Oncology, Department of Internal Medicine, Chang Gung Memorial Hospital at Linkou
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Background] Hsieh JC, Lin HC, Huang CY, Hsu HL, Wu TM, Lee CL, Chen MC, Wang HM, Tseng CP. Prognostic value of circulating tumor cells with podoplanin expression in patients with locally advanced or metastatic head and neck squamous cell carcinoma. Head Neck. 2015 Oct;37(10):1448-55. doi: 10.1002/hed.23779. Epub 2014 Jul 24. PMID 24844673
- [Background] Huang SB, Wu MH, Lin YH, Hsieh CH, Yang CL, Lin HC, Tseng CP, Lee GB. High-purity and label-free isolation of circulating tumor cells (CTCs) in a microfluidic platform by using optically-induced-dielectrophoretic (ODEP) force. Lab Chip. 2013 Apr 7;13(7):1371-83. doi: 10.1039/c3lc41256c. PMID 23389102
- [Background] Huang SB, Wang SS, Hsieh CH, Lin YC, Lai CS, Wu MH. An integrated microfluidic cell culture system for high-throughput perfusion three-dimensional cell culture-based assays: effect of cell culture model on the results of chemosensitivity assays. Lab Chip. 2013 Mar 21;13(6):1133-43. doi: 10.1039/c2lc41264k. PMID 23353927